CLINICAL TRIAL: NCT07055711
Title: Association Between Work-Related Stress and Peripheral Neuropathic Pain in Female Breast Cancer Survivors Post-Chemotherapy
Brief Title: Association Between Work-Related Stress and Peripheral Neuropathic Pain in Female Breast Cancer Post CT
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: DPT/Batch-Fall20/1016
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Peripheral Neuropathic Pain — to find out the association between work-related stress and peripheral neuropathic pain in female breast cancer survivors post-chemotherapy.

SUMMARY:
This research aims to find the association between work-related stress and peripheral neuropathic pain in female breast cancer survivors post-chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Females who have completed chemotherapy at least o1 year prior to study.
* Aged 29-51.
* Females who is currently employed.
* Females who have done chemotherapy for stage 1,2,3.
* Females who underwent chemotherapy cycles 6-8.
* Females who are willing to participate in the study

Exclusion Criteria:

* Females suffering from psychiatric conditions such as anxiety and depression.
* Females suffering from diabetes.
* Females who have active cancer.
* Females with mastectomy.
* Absent from treatment for more than 2 weeks will be excluded from the study.

Ages: 21 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: to find out the Association Between Work-Related Stress and Peripheral Neuropathic Pain in Female Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Douleur Neuropathique 4 (DN4) Questionnaire | 6 Month
  The DN4 questionnaire is used to assess the neuropathic pain, if the score is > 4 it indicates the neuropathic pain is present while <3 than is unlikely.
visual analog scale | 6 Months
  The visual analog scale provide quantitative measurement of pain level which is from no pain to severe pain . The range of the scale is in between 0-10mm. 0-4 is consider as no pain, 5-44 is consider as mild pain,45-74 is moderate and > 75 is consider as severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore City, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No